CLINICAL TRIAL: NCT03203720
Title: Brief Motivational Intervention to Improve Medication Adherence for Adolescents With Bipolar Disorder
Acronym: BMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Tina R Goldstein, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH092424
Record Dates: First submitted 2017-06-23; First posted 2017-06-29 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder; Medication Adherence
Keywords: adherence; adolescent; Motivational Intervention
MeSH Terms: conditions — Bipolar Disorder; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Randomized trial comparing Brief Motivational Intervention + Standard Care versus Standard Care Alone
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors blind to treatment group of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (SC) (No Intervention): Standard Care (SC) in a specialty mood disorders clinic for youth with mood disorders.
- SC + Brief Motivational Intervention (Experimental): Standard Care (SC) in a specialty mood disorders clinic plus a Brief Motivational Intervention (BMI) targeting medication adherence.
  Interventions: Behavioral: Brief Motivational Intervention

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — A brief motivational intervention centered around Motivational Interviewing (MI) techniques. Sessions are adjunct to standard clinical care, and focus on psychoeducation regarding treatment for bipolar disorder, and resolving ambivalence regarding taking medications for mood disorder.
  Other Names: BMI
  Arms: SC + Brief Motivational Intervention

SUMMARY:
Adolescence is the peak onset period for serious and persistent psychiatric disorders. Treatment guidelines for management of major psychiatric disorders in youth include pharmacotherapy. There has been substantial progress in recent years in identifying effective medications for youth with psychiatric disorders. However, adherence to prescribed medications among psychiatric populations is notoriously low, and adolescents rank among the least adherent of all patient populations. Given that the consequences of poor medication adherence among youth with chronic mental illness are far-reaching, including hospitalization, poor functioning, and suicide, there is a desperate need for interventions targeting medication adherence in this population.

DETAILED DESCRIPTION:
Adolescence is the peak period of onset for serious and persistent psychiatric disorders. Treatment guidelines for the management of major psychiatric disorders in adolescence indicate pharmacotherapy is a critical element of effective treatment. Unfortunately, adolescence is a particularly vulnerable window for poor medication adherence, and little is known about the timecourse and specific factors associated with poor medication adherence in this population. Given that the consequences of poor medication adherence among youth with chronic mental illness are far-reaching, and include hospitalization, profound functional impairment and even suicide, there is a desperate need for interventions targeting medication adherence in this population. Motivational Interviewing (MI) is an evidence-based approach focused on enhancing motivation for change. This model holds great promise for improving medication adherence in adolescents with psychiatric disorders because it is developmentally sensitive, acceptable to patients and providers, and readily disseminable across clinical settings. Research demonstrates that brief motivational interventions (BMIs) utilizing a MI approach result in improved treatment adherence among youth with a variety of chronic medical conditions. Although widely applied for adolescent substance use behaviors, BMIs have yet to be examined for improving medication adherence in youth with severe psychiatric disorders. Adolescents with bipolar disorder (BP) are an ideal population with whom to develop a BMI for medication adherence because adolescents with BP are among the least adherent of any psychiatric population. Experience developing a BMI for this challenging population will directly inform intervention for youth with a range of chronic psychiatric disorders. The purpose of the proposed study is to conduct a small randomized trial comparing CABS Standard Care (SC) augmented with the BMI versus SC alone. Outcomes will be assessed monthly over 6 months. Participants will include 40 adolescents with BP. This approach is in direct accord with the National Institute of Mental Health (NIMH) Strategic Plan in which the development and testing of innovative interventions to reduce risk and positively alter trajectories of mental illness are informed by research findings regarding robust and malleable risk factors. Research in this area is of great public health importance, as it has the potential to lessen costs, disrupt the cycle of poor outcomes, and minimize the long-term debilitating effects of these serious disorders.

ELIGIBILITY:
Inclusion Criteria:

1. age 12 years, 0 months to 22 years, 11 months;
2. a diagnosis of BP spectrum disorder via semi-structured interview;
3. willing to engage in treatment at the BP specialty clinic;
4. English fluency and understanding, as the study consists of interviews and surveys that necessitate English fluency and understanding;
5. able and willing to give informed consent/assent to participate.

Exclusion Criteria:

1. evidence of mental retardation, pervasive developmental disorder, or organic central nervous system disorder by semi-structured interview, parent report, medical history, or school records;
2. a life-threatening medical condition requiring immediate treatment;
3. current victim of sexual or physical abuse.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Objective Medication Adherence | 6 months
  Medication adherence via electronic pillbox
Subjective Medication Adherence | 6 months
  Self-reported medication adherence

SECONDARY OUTCOMES:
Mood disorder symptoms | Quarterly over 6 months
  Depressive and manic symptoms as measured via semi-structured interview

CONTACTS AND LOCATIONS:
Overall Officials: Tina R Goldstein, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstein TR, Krantz ML, Fersch-Podrat RK, Hotkowski NJ, Merranko J, Sobel L, Axelson D, Birmaher B, Douaihy A. A brief motivational intervention for enhancing medication adherence for adolescents with bipolar disorder: A pilot randomized trial. J Affect Disord. 2020 Mar 15;265:1-9. doi: 10.1016/j.jad.2020.01.015. Epub 2020 Jan 7. PMID 31957686